CLINICAL TRIAL: NCT06042426
Title: Effects of Perioperative Intravenous Dexamethasone in Clinical Outcomes After Total Knee Arthroplasty in a Hispanic Population: A Randomized Controlled Trial
Brief Title: Effects of Perioperative Intravenous Dexamethasone in Clinical Outcomes After Total Knee Arthroplasty in a Hispanic Population
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2306117408
Record Dates: First submitted 2023-08-03; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis, Knee
Keywords: TKA; Primary osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Dexamethasone; Morphine; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients receiving intravenous dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone
- Patients receiving intravenous morphine and oral oxycodone (Active Comparator)
  Interventions: Drug: Morphine; Drug: Oxycodone and acetaminophen

INTERVENTIONS:
Drug: Dexamethasone — Two 8 mg doses. One dose applied prior to incision and the other at POD1
  Arms: Patients receiving intravenous dexamethasone
Drug: Morphine — Morphine 0.1 mg per kg intravenous every 6 hours
  Arms: Patients receiving intravenous morphine and oral oxycodone
Drug: Oxycodone and acetaminophen — 2 tabs of oral oxycodone combined with acetaminophen every 6 hours (the same pill includes both drugs)
  Arms: Patients receiving intravenous morphine and oral oxycodone

SUMMARY:
The purpose of this study is to evaluate the efficacy of an intravenous (IV) perioperative dexamethasone regime in the clinical outcomes after a robotic-assisted Total Knee Arthroplasty (TKA) in a Hispanic population. The study aims to propose an alternative to opioid-based pain treatment following TKA. The study hopefully validates the use of a two-dose, 8mg intravenous dexamethasone regimen for improving pain and range of motion scores in patients undergoing primary, unilateral TKA for osteoarthritis. One dose will be applied prior to incision and the other at post-operative day (POD) 1.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Hispanic self-identification
* Primary robotic-assisted TKA for treatment of primary osteoarthritis
* Age ≥ 21
* Receiving seven days of inpatient rehabilitation after medical discharge
* Patient with adequate glycemic control (HbA1c<7.5%)
* Patients who provide written informed consent

Exclusion Criteria:

* Age ≤ 21
* Chronic steroid use prior to surgery
* Previous allergies or adverse reactions to steroid drugs
* Indications for surgery other than primary osteoarthritis
* History of narcotics abuse such as opioids
* Surgeries performed without robotic-assistance
* Outpatient or Home rehabilitation programs after medical discharge
* Requirement of revision surgery orthopaedic implants
* Patients with inadequate glycemic control (HbA1c≥7.5%)
* Other medical conditions, such as osteoporosis, fungal infections, glaucoma, joint infections, peptic ulcer disease which could worsen with steroid administration.

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
POD 1 Visual Analogue Scale Pain Scores | Measured at 7:00AM day after surgery
  Range: 0-10 (10 indicates highest degree of pain)
POD 2 Visual Analogue Scale Pain Scores | Measured at 7:00AM two days after surgery
  Range: 0-10 (10 indicates highest degree of pain)
POD 3 Visual Analogue Scale Pain Scores | Measured at 7:00AM three days after surgery
  Range: 0-10 (10 indicates highest degree of pain)
POD 1 Range of Motion | Measured at 7:00AM the day after surgery
POD 2 Range of Motion | Measured at 7:00AM two days after surgery
POD 3 Range of Motion | Measured at 7:00AM three days after surgery

SECONDARY OUTCOMES:
Daily Dextrose Concentration (mg/dL) | Measured at 7:00AM for 3 days after surgery
Length of Stay | From hospital admission to the date of discharge (About 3 days)
  Measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Antonio M López Otero, MD, Principal Investigator — Orthopaedic Surgery Section, University of Puerto Rico Medical Sciences Campus San Juan, Puerto Rico
Locations (1):
- University of Puerto Ric-Dr. Federico Trilla Hospital, Carolina, Puerto Rico